CLINICAL TRIAL: NCT03016962
Title: Usefulness of Cap-assisted Colonoscopy in Patients With Prior Abdominal Surgery: A Randomized, Controlled Trial
Brief Title: Usefulness of Cap-assisted Colonoscopy in Patients With Prior Abdominal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Jeong-Seon Ji, Dr, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Cap
Record Dates: First submitted 2017-01-09; First posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Insertion Time

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cap-assisted colonoscopy (Experimental): cap-assisted colonoscopy
  Interventions: Device: cap-assisted colonoscopy
- Standard colonoscopy (Active Comparator): Standard colonoscopy
  Interventions: Device: Standard colonoscopy

INTERVENTIONS:
Device: cap-assisted colonoscopy — cap-assisted colonoscopy
  Arms: Cap-assisted colonoscopy
Device: Standard colonoscopy — Standard colonoscopy
  Arms: Standard colonoscopy

SUMMARY:
The potential benefit of using the cap is that it helps in luminal orientation at bends by keeping the colonic mucosa away from the lens at the colonoscope tip. Colonoscopy in patients with a history of abdominal surgery is considered to be difficult due to adhesion-related bowel angulations. There were few study evaluating usefulness of cap-assisted colonoscopy in patients with prior abdominal surgery. The investigators designed a randomized, controlled trial to verify the usefulness of cap-assisted colonoscopy in patients with prior abdominal surgery.

DETAILED DESCRIPTION:
The potential benefit of using the cap is that it helps in luminal orientation at bends by keeping the colonic mucosa away from the lens at the colonoscope tip. This assists in negotiating sharp turns by better anticipation of the direction. Cap-assisted colonoscopy can be tried as a salvage procedure in cases of failed cecal intubation with regular colonoscopy. Colonoscopy in patients with a history of abdominal surgery is considered to be difficult due to adhesion-related bowel angulations. There were few study evaluating usefulness of cap-assisted colonoscopy in patients with prior abdominal surgery. The investigators designed a randomized, controlled trial to verify the usefulness of cap-assisted colonoscopy in patients with prior abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with history of abdominal or pelvic surgery

Exclusion Criteria:

* Previous colorectal resection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1046 (Estimated)
Dates: Start 2017-02; Primary Completion 2020-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Insertion time | Day 1

SECONDARY OUTCOMES:
Patient discomfort | Day 1
  10-point visual analog scale
Overall technical ease | Day 1
  10-point visual analog scale

IPD SHARING:
Plan to Share IPD: No